CLINICAL TRIAL: NCT00686842
Title: A Phase I/II Trial of PTC299 in Patients With HIV-Related Kaposi's Sarcoma
Brief Title: PTC299 in Treating Patients With HIV-Related Kaposi Sarcoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Drug supply unavailable.
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH); PTC Therapeutics (Industry); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC-059; U01CA121947 (NIH); CDR0000596565 (Other: NCI); PTC299-ONC-005-KS (Other: PTC Therapeutics)
Record Dates: First submitted 2008-05-29; First posted 2008-05-30 (Estimated); Results first posted 2012-03-05 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Kaposi's Sarcoma
Keywords: HIV infection; AIDS-related Kaposi sarcoma; recurrent Kaposi sarcoma; Treatment Experienced
MeSH Terms: conditions — Sarcoma, Kaposi; HIV Infections; AIDS-related Kaposi sarcoma | interventions — emvododstat; Gene Expression Profiling; Polymerase Chain Reaction; Immunohistochemistry; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VEGF Inhibitor PTC299 (Experimental): Single arm study - all subjects received PTC299
  Interventions: Drug: VEGF inhibitor PTC299; Genetic: gene expression analysis; Genetic: polymerase chain reaction; Genetic: protein expression analysis; Other: immunohistochemistry staining method; Other: laboratory biomarker analysis; Other: pharmacological study; Procedure: biopsy

INTERVENTIONS:
Drug: VEGF inhibitor PTC299 — 20 mg capsules to be taken by mouth BID. Three dose levels will be evaluated: 40 mg, 80mg, and 100mg BID. Subjects will receive PTC299 in consecutive 28-day cycles for a maximum of 12 cycles.
Genetic: gene expression analysis — To describe the effects of PTC299 on viral gene expression and cellular gene transcription in KS tumor biopsies using real-time QPCR-based profiling.
Genetic: polymerase chain reaction — To describe the effects of PTC299 on viral gene expression and cellular gene transcription in KS tumor biopsies using real-time QPCR-based profiling.
Genetic: protein expression analysis — To describe the effects of PTC299 on viral gene expression and cellular gene transcription in KS tumor biopsies using real-time QPCR-based profiling.
Other: immunohistochemistry staining method — To describe the effects of PTC299 on KS tumor biopsies with respect to expression of VEGF, the VEGFR-2 and -3, phospho-Akt, p53, HIF-1α and proliferation, measured by Ki-67 staining.
Other: laboratory biomarker analysis — To describe the effects of PTC299 on KS tumor biopsies with respect to expression of VEGF, the VEGFR-2 and -3, phospho-Akt, p53, HIF-1α and proliferation, measured by Ki-67 staining.
Other: pharmacological study — To describe the pharmacokinetics of PTC299 in patients with HIV-associated KS. To describe the effects of PTC299 on circulating VEGF, VEGFR and cytokine levels in patients with HIV-associated KS.
Procedure: biopsy — To describe the effects of PTC299 on KS tumor biopsies with respect to expression of VEGF, the VEGFR-2 and -3, phospho-Akt, p53, HIF-1α and proliferation, measured by Ki-67 staining.

SUMMARY:
RATIONALE: PTC299 may stop the growth of Kaposi sarcoma by blocking blood flow to the tumor.

PURPOSE: This phase I/II trial is studying the side effects and best dose of PTC299 and to see how well it works in treating patients with HIV-related Kaposi sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To define the safety and toxicity of anti-VEGF small molecule PTC299 in patients with HIV-related Kaposi sarcoma.
* To establish the maximum tolerated dose of this drug in these patients.
* To estimate the response rate in patients treated with this drug.

Secondary

* To describe the pharmacokinetics of this drug in these patients.
* To describe the effects of this drug on serum and plasma VEGF, VEGFR, and cytokine profiles in these patients.
* To describe the effects of this drug on HIV and KSHV viral loads in these patients.
* To describe the effects of this drug on T-lymphocyte subsets (i.e., CD4 and CD8) in these patients.
* To describe the effects of this drug on VEGF, VEGFR-2 and -3, phospho-Akt, p53, and HIF-1α expression and tumor cell proliferation, as measured by Ki-67 staining, in tumor biopsy samples obtained from these patients.
* To describe the effects of this drug on viral gene expression and cellular gene transcription, as measured by real-time quantitative PCR-based profiling, in tumor biopsy samples obtained from these patients.

OUTLINE: This is a multicenter, phase I dose-escalation study of anti-VEGF small molecule PTC299 followed by a phase II study.

Patients receive oral anti-VEGF small molecule PTC299 twice daily on days 1-28. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity. Patients who do not demonstrate an objective response of their Kaposi sarcoma (KS) lesions after 6 courses of treatment are removed from the study.

Patients undergo blood sample collection and punch biopsies periodically during study for correlative laboratory studies. Biopsy samples are assessed for VEGF, VEGFR-2, VEGFR-3, phospho-Akt, KSHV LANA, orf59, p53, and HIF-1α expression by IHC; tumor cell proliferation by Ki-67 staining; and viral gene expression at the messenger RNA level and KSHV transcription by real-time quantitative PCR-based profiling. Blood samples are assessed for pharmacokinetics and levels of secreted cytokines or other potential serum markers characteristic for KS.

After completion of study treatment, patients are followed at 30 days.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Biopsy-proven Kaposi sarcoma (KS) involving the skin (with or without lymph node), oral cavity, gastrointestinal (GI) tract, and/or lung

  * Patients with GI and/or pulmonary involvement must be asymptomatic or minimally symptomatic and not require systemic cytotoxic chemotherapy
* Has at least five bidimensionally measurable cutaneous lesions that have not been previously irradiated AND can be used as indicator lesions

  * Must have a sufficient number of non-indicator cutaneous lesions measuring ≥ 4 x 4 mm available to obtain a total of four 3-mm punch biopsies (two at baseline and two during the course of study treatment)
* Serologic documentation of HIV infection, as evidenced by positive ELISA, western blot, or other federally approved licensed HIV test OR a detectable blood level of HIV RNA
* Patients receiving antiretroviral therapy for HIV infection are eligible provided they have been on a stable regimen for ≥ 12 weeks prior to study entry AND there is no evidence of improvement in KS during those 12 weeks or there is evidence of progression of KS within the immediate 4 weeks prior to study entry
* No symptomatic visceral KS requiring cytotoxic therapy

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* Life expectancy ≥ 3 months
* Absolute neutrophil count ≥ 1,000/mm³
* Platelet count ≥ 75,000/mm³
* Hemoglobin ≥ 8 g/dL
* Creatinine ≤ 2.0 mg/dL
* Total bilirubin normal (grade 0)

  * No specific limit of total serum bilirubin for patient receiveing indinavir or atazanavir therapy AND direct serum bilirubin ≤ 30% of total bilirubin
* AST and ALT ≤ 2.5 times upper limit of normal (grade 1)
* INR and aPTT normal
* Proteinuria < 2+
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for up to 3 months after completion of study treatment
* Capable of complying with the study, in the opinion of the investigator
* No acute, active opportunistic infection (other than oral thrush or genital herpes) within the past 14 days
* No other concurrent neoplasia requiring cytotoxic therapy
* No history of any of the following:

  * Myocardial infarction
  * Severe/unstable angina
  * Coronary/peripheral artery bypass graft
  * Symptomatic congestive heart failure
  * Cerebrovascular accident
  * Transient ischemic attack
  * Pulmonary embolism
  * Deep vein thrombosis
  * Other significant thromboembolic event
* No known coagulopathy or bleeding diathesis
* No history of CNS, pulmonary, GI, or urinary bleeding
* No known history of drug-induced liver injury
* Resting systolic blood pressure ≤ 160 mm Hg or diastolic blood pressure ≤ 100 mm Hg
* No history of or ongoing clinically significant illness, medical condition, surgical history, physical finding, ECG finding, or laboratory abnormality that, in the opinion of the investigator, could affect the safety of the patient, alter the absorption of the study drug, or impair the assessment of study results

PRIOR CONCURRENT THERAPY:

* More than 4 weeks since prior and no other concurrent anti-neoplastic therapy for KS, including chemotherapy, radiotherapy, local therapy, or biological therapy
* More than 60 days since prior local therapy for any KS-indicator lesion unless the lesion has clearly progressed since treatment

  * Any prior local therapy for indicator lesions (regardless of the elapsed time) should not be allowed unless there is evidence of clear-cut progression of that lesion
* More than 28 days since prior and no other concurrent investigational drugs or therapy (other than antiretroviral therapy or agents available on a treatment IND)
* More than 30 days since prior major surgery and recovered
* More than 14 days since prior treatment for an acute infection (other than oral thrush or genital herpes) or other serious medical illness
* No concurrent surgical procedures
* No concurrent systemic corticosteroid therapy, other than replacement doses
* No concurrent anticoagulant therapy, including warfarin, heparin (including low molecular weight heparin), or antiplatelet drugs (e.g., clopidogrel bisulfate)

  * Concurrent aspirin or nonsteroidal anti-inflammatory drugs (NSAIDs) allowed provided the dose does not exceed the maximum recommended dose

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-09; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan E. Krown, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - UCLA Clinical AIDS Research and Education (CARE) Center, Los Angeles, California
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Floyd and Delores Jones Cancer Institute at Virginia Mason Medical Center, Seattle, Washington

REFERENCES:
- [Background] Bender Ignacio RA, Lee JY, Rudek MA, Dittmer DP, Ambinder RF, Krown SE; AIDS Malignancy Consortium (AMC)-059 Study Team. Brief Report: A Phase 1b/Pharmacokinetic Trial of PTC299, a Novel PostTranscriptional VEGF Inhibitor, for AIDS-Related Kaposi's Sarcoma: AIDS Malignancy Consortium Trial 059. J Acquir Immune Defic Syndr. 2016 May 1;72(1):52-7. doi: 10.1097/QAI.0000000000000918. PMID 26689971

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | VEGF Inhibitor PTC299
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | VEGF Inhibitor PTC299
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.7 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Safety and Toxicity of Anti-VEGF Small Molecule PTC299
Description: Patients who experienced an adverse event of grade 3 or greater
Time Frame: All study visits
Measure: Number; unit: participants
Arm/Group | VEGF Inhibitor PTC299
Number analyzed (Participants) | 17
participants | 7

2. Primary Outcome: Maximum Tolerated Dose
Time Frame: After each group of 3 subjects completes cycle 1 of treatment
Reporting Status: Not Posted

3. Primary Outcome: Response to Treatment
Time Frame: After each 28-day cycle of treatment and at discontinuation of therapy
Reporting Status: Not Posted

4. Secondary Outcome: Pharmacokinetics
Time Frame: Days 1, 15, 28, 57
Reporting Status: Not Posted

5. Secondary Outcome: Effects of Study Drug on Serum and Plasma VEGF, VEGFR, and Cytokine Profiles
Time Frame: On the first day of every 28-day cycle of treatment, Day 15, and treatment discontinuation
Reporting Status: Not Posted

6. Secondary Outcome: Effects of Study Drug on HIV and KSHV Viral Loads
Time Frame: Screening, end of cycle 1, end of every third cycle thereafter, and treatment discontinuation
Reporting Status: Not Posted

7. Secondary Outcome: Effects of Study Drug on T-lymphocyte Subsets (i.e., CD4 and CD8)
Time Frame: Screening, day 29, every 3 cycles thereafter, and at treatment discontinuation
Reporting Status: Not Posted

8. Secondary Outcome: Effects of Study Drug on VEGF, VEGFR-2 and -3, Phospho-Akt, p53, and HIF-1α Expression and Tumor Cell Proliferation, as Measured by Ki-67 Staining, in Tumor Biopsy Samples
Time Frame: Screening and day 28
Reporting Status: Not Posted

9. Secondary Outcome: Effects of Study Drug on Viral Gene Expression and Cellular Gene Transcription, as Measured by Real-time Quantitative PCR-based Profiling, in Tumor Biopsy Samples
Time Frame: Screening and day 28
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | VEGF Inhibitor PTC299
Serious Adverse Events (participants affected / at risk) | 3/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VEGF Inhibitor PTC299 (N=17)
Sudden death (General disorders) | 1 (1)
Renal and urinary disorder (Renal and urinary disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VEGF Inhibitor PTC299 (N=17)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Acidosis (General disorders) | 2 (2)
alanine aminotransferase increases (Metabolism and nutrition disorders) | 2 (4)
alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Arthralgia (Immune system disorders) | 2 (2)
Blood bilirubin increased (Investigations) | 3 (3)
Cholesterol high (Infections and infestations) | 4 (6)
Constipation (Gastrointestinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Creatinine increased (Investigations) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 4 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Edema face (General disorders) | 2 (2)
Edema limbs (General disorders) | 3 (3)
Fatigue (General disorders) | 5 (6)
Headache (Nervous system disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (8)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 5 (6)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (5)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 7 (10)
Neutrophil count decreases (Blood and lymphatic system disorders) | 2 (2)
Pain (Musculoskeletal and connective tissue disorders) | 5 (6)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Proteinuria (Renal and urinary disorders) | 3 (4)
Skin and subcutaneous tissue disorder (Skin and subcutaneous tissue disorders) | 2 (2)
Skin infection (Infections and infestations) | 3 (4)
Vomiting (Gastrointestinal disorders) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2010-10-22): https://cdn.clinicaltrials.gov/large-docs/42/NCT00686842/Prot_SAP_001.pdf